CLINICAL TRIAL: NCT06855069
Title: A Multi-center, Randomized, Open-label, Controlled, Phase III Clinical Study Evaluating HS-20089 vs. Investigator's Choice of Chemotherapy in the Treatment of Platinum-resistant Recurrent Epithelial Ovarian Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Brief Title: HS-20089 for Injection in Patients With Platinum-Resistant Recurrent Epithelial Ovarian Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-20089-301
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer
Keywords: Platinum-resistant recurrent epithelial ovarian cancer; HS-20089; randomized; phase III
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment group 1: HS-20089 (Experimental)
  Interventions: Drug: HS-20089
- Treatment group 2: Investigator's choice of chemotherapy (Active Comparator)
  Interventions: Drug: Paclitaxel; Drug: Doxorubicin; Drug: Topotecan

INTERVENTIONS:
Drug: HS-20089 — HS-20089 dose 1
  Arms: Treatment group 1: HS-20089
Drug: Paclitaxel — Paclitaxel dose 2
  Arms: Treatment group 2: Investigator's choice of chemotherapy
Drug: Doxorubicin — Doxorubicin dose 3
  Arms: Treatment group 2: Investigator's choice of chemotherapy
Drug: Topotecan — Topotecan dose 4
  Arms: Treatment group 2: Investigator's choice of chemotherapy

SUMMARY:
This study is a randomized, open-label, controlled, phase III study to evaluate the efficacy and safety of HS-20089 versus investigator's choice of chemotherapy in patients with platinum-resistant recurrent epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent.
2. 18 years and older, female.
3. Pathologically diagnosed epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.
4. Patients must have platinum-resistant disease
5. Be able to provide fresh or archived tumor tissue.
6. At least one measurable lesion according to RECIST v1.1.
7. Eastern Cooperative Oncology Group (ECOG) score: 0-1.
8. With a life expectancy > 12 weeks.
9. Adequate bone marrow reserve and organ function.
10. Contraception is required during the trial.

Exclusion Criteria:

1. Prior treated with TOP1 inhibitors or ADCs with TOP1 inhibitors as payload.
2. Previous or co-existing malignancies.
3. Uncontrolled pleural effusion, pericardial effusion, or abdominal effusion requiring clinical intervention.
4. Received systemic anticancer treatments 4 weeks prior to the initiation of the study treatment.
5. Unresolved CTCAE ≥grade 2 toxicities from previous anticancer therapy.
6. History of severe hypersensitivity reactions to either the drug substances or inactive ingredients of HS-20089.
7. Any serious or uncontrolled medical disorder in the opinion of the investigator that may increase the risk associated with the study participation or study drug administration.
8. Other inappropriate situation considered by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-03-07 (Estimated); Study Completion 2029-03-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) assessed by Blinded Independ Review Committee (BIRC) as per RECIST 1.1 | Screening up to study completion, an average of 1 year

SECONDARY OUTCOMES:
Overall Survival (OS) | Screening up to study completion, an average of 1 year
Objective Response Rate (ORR), assessed by site investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Duration of Response (DoR), assessed by site investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Disease Control Rate (DCR), assessed by site investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Objective Response Rate (ORR), assessed by BIRC as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Duration of Response (DoR), assessed by BIRC as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Disease Control Rate (DCR), assessed by BIRC as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Adverse Events | Screening up to study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China